CLINICAL TRIAL: NCT03577223
Title: Egg Effects on the Immunomodulatory Properties of HDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fairfield University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Catherine Andersen, Associate Professor of Biology, Fairfield University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0511
Record Dates: First submitted 2018-06-15; First posted 2018-07-05 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Lipid Metabolism; Inflammation
Keywords: Egg; HDL; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole Eggs (Experimental)
  Interventions: Other: Whole Eggs
- Egg White-Based Egg Substitute (Active Comparator)
  Interventions: Other: Egg White-Based Egg Substitute

INTERVENTIONS:
Other: Whole Eggs — 3 whole eggs per day for 4 weeks
  Arms: Whole Eggs
Other: Egg White-Based Egg Substitute — 3-egg equivalent of egg white-based egg substitute per day for 4 weeks
  Arms: Egg White-Based Egg Substitute

SUMMARY:
The purpose of this study is to investigate the effects of egg intake on markers of HDL function and immune inflammation in healthy adults.

DETAILED DESCRIPTION:
28 healthy men and women (age 18-35 years old) will be recruited to participate in a 16-week randomized crossover study. Upon enrollment, all subjects will enter a 4-week run-in egg-free period where they will refrain from consuming any egg-based foods (Period 1). Subjects will then enter the first intervention period, where they be randomly assigned to consume either 3 whole eggs/day or the equivalent amount of egg white-based egg substitute/day for 4 weeks (Period 2). Afterwards, subjects will enter a 4-week washout period where egg-based foods are restricted (Period 3), followed by a second intervention period, where they be assigned to the alternative whole egg- or egg white-based treatment for 4 weeks (Period 4). Subjects will come to the Department of Biology at Fairfield University every two weeks to check-in, and to pick up their egg products during the intervention periods. Subjects will be asked to maintain their normal diet and physical activity practices throughout all periods of the study. Subjects will complete 5-day dietary records and physical activity logs at the end of each study period.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* Body mass index (BMI) < 30 kg/m2, or < 30% body fat for men and < 40% body fat for women
* Willingness to consume eggs or egg whites on a daily basis during study periods

Exclusion Criteria:

* < 18 years old; > 35 years old
* BMI ≥ 30 kg/m2, or ≥ 30% body fat for men and ≥ 40% body fat for women
* Self-reported history of diabetes mellitus, coronary heart disease, stroke, renal problems, liver disease, cancer, pregnancy or lactation, autoimmunity, chronic infections, or egg allergy
* Taking lipid-lowering medications (e.g. statins, fibrates)
* A preexisting medical condition or implanted medical device that prevents participation in bioelectrical impedance measurements of body composition
* Clinical lipid and glucose values that are highly elevated, including fasting triglycerides levels higher than 500 mg/dL, fasting glucose higher than 126 mg/dL, and plasma total cholesterol greater than 240 mg/dL

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Fasted HDL-cholesterol | 16 weeks
  Measurement of fasted plasma HDL-cholesterol levels (mg/dL) at the end of the run-in period, and two intervention arms.

SECONDARY OUTCOMES:
Fasted HDL lipid composition | 16 weeks
  HDL subfractions (d = 1.063-1.21) will be isolated from plasma by ultracentrifugation collected at the end of the run-in period and two intervention arms. HDL fractions will be analyzed for glycerphospholipid (phosphatidylcholine, phosphatidylethanolamine, lysophosphatidylcholine, phosphatidylinositol) and sphingolipid (sphingomyelin) composition by mass spectrometry. Each lipid class will be presented as a percent (%) of total HDL lipids.
Cholesterol-accepting capacity of serum | 16 weeks
  The cholesterol efflux from macrophages to subject serum will be measured at the end of the egg-free run-in period and both intervention periods using a fluorescent cholesterol efflux kit. Results will be expressed as % cholesterol efflux, calculated as (fluorescence intensity of media/[fluorescent intensity of cell lysates + media]) x 100.
Inflammatory potential of peripheral blood mononuclear cells | 16 weeks
  Peripheral blood mononuclear cells (PBMCs) will be isolated at the end of the egg-free run-in period and both intervention periods. PBMCs will be cultured ex vivo and stimulated with lipopolysaccharide. Media will be collected to measure tumor necrosis factor alpha concentrations (pg/mL) in cell media.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J Andersen, PhD, RD, Principal Investigator — Fairfield University
Locations (1):
- Fairfield University, Fairfield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No